CLINICAL TRIAL: NCT04310462
Title: A Quality Improvement Study to Measure the Effectiveness of an E-prescribing Interface to Reduce Dosage of Hydroxychloroquine Above Current Guidelines
Brief Title: Effectiveness of an EHR Interface to Reduce Dosage of Hydroxychloroquine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study investigators became aware of an internal error that overrode randomization of providers; therefore, the study randomization for this study was no longer present.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCSF-16-21347
Record Dates: First submitted 2020-01-21; First posted 2020-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New eRX Interface (Experimental): Providers assigned to the intervention arm will be presented with a new eRX interface upon writing new prescriptions for hydroxychloroquine in the EHR.
  Interventions: Other: New e-prescribing interface
- Standard Interface (No Intervention): Providers assigned to the no intervention arm will be presented with the usual ordering interface when prescribing new prescriptions for hydroxychloroquine in the EHR.

INTERVENTIONS:
Other: New e-prescribing interface — The goal of this study is to conduct a pragmatic trial to assess the utility of a new e-prescribing (eRX) interface for prescriptions of hydroxychloroquine (HCQ). Through randomization of clinicians to the new interface, the investigators will measure the effectiveness of the system in reducing the number of individuals prescribed HCQ over current guidelines.
  Arms: New eRX Interface

SUMMARY:
Hydroxychloroquine (HCQ) is a disease-modifying, anti-rheumatic drug that regulates immune system activity and is typically prescribed to treat rheumatoid arthritis and systemic lupus erythematosus, as well as other immune conditions. Although generally well tolerated, study data have demonstrated that long-term use of HCQ may lead to irreversible and potentially vision-threatening retinal toxicity. The American Academy of Ophthalmology (AAO) issued guidelines in 2011, and again in 2016 that recommended dosing of HCQ be based on an individual's body weight, and also outlined how and when to screen for retinal toxicity. While clinicians have been aware of the potential side effects of HCQ for decades, studies have shown that many patients continue to receive higher than recommended doses.

The goal of this study is to conduct a pragmatic trial to assess the utility of a new e-prescribing (eRX) interface for prescriptions of hydroxychloroquine (HCQ). The investigators will measure the effectiveness of the system in reducing the number of individuals prescribed HCQ over current guidelines by randomizing clinicians to the new interface. Ideally, the eRX interface will result in a lower number of potential adverse events (i.e. retinal toxicity) associated with high-dose, long-term use of HCQ.

ELIGIBILITY:
Inclusion Criteria:

* All providers that prescribed hydroxychloroquine in the year previous to the intervention start date in rheumatology and dermatology clinics

Exclusion Criteria:

* Inactive providers in rheumatology and dermatology clinics

Max Age: 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of dosage above guidelines: 6.5 mg/kg (2011) | Post intervention: 1 year
  Prevalence of dosage above 6.5 mg/kg
Prevalence of dosage above guidelines: 6.5 mg/kg (2011) | Post intervention: 2 years
  Prevalence of dosage above 6.5 mg/kg
Prevalence of dosage above guidelines: 6.5 mg/kg (2011) | Post intervention: 3 years
  Prevalence of dosage above 6.5 mg/kg
Prevalence of dosage above guidelines: 5.0 mg/kg (2016) | Post intervention: 1 year
  Prevalence of dosage above 5.0 mg/kg
Prevalence of dosage above guidelines: 5.0 mg/kg (2016) | Post intervention: 2 years
  Prevalence of dosage above 5.0 mg/kg
Prevalence of dosage above guidelines: 5.0 mg/kg (2016) | Post intervention: 3 years
  Prevalence of dosage above 5.0 mg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Jinoos Yazdany, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Summary level data may be provided upon request